CLINICAL TRIAL: NCT02146937
Title: A Phase 2 Study of Bicalutamide Plus Finasteride in Men With MRI Detectable Prostate Nodules Undergoing Active Surveillance
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to lack of accrual for this study. PI decided to close the study.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1408; NA_00092522 (Other: JHMIRB)
Record Dates: First submitted 2014-05-01; First posted 2014-05-26 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Detectable Prostate Nodules
Keywords: active surveillance; MRI/transrectal ultrasound fusion guided biopsy; biopsy
MeSH Terms: interventions — bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination therapy- bicalutamide and finasteride (Experimental): 3-month (90-day) course of bicalutamide 50 mg by mouth daily and finasteride 5 mg by mouth daily
  Interventions: Drug: Bicalutamide plus Finasteride- Combination therapy

INTERVENTIONS:
Drug: Bicalutamide plus Finasteride- Combination therapy — 3-month (90-day) course of bicalutamide 50 mg by mouth daily and finasteride 5 mg by mouth daily

SUMMARY:
This is an open label, single site, single arm Phase II study to evaluate the combination of bicalutamide plus finasteride in men with MRI detectable significant prostate nodules followed on active surveillance.

DETAILED DESCRIPTION:
This research is being done to determine the negative re-biopsy rate as determined by MRI/TRUS fusion guided biopsy targeting the dominant nodule site defined by pre-treatment MRI following three months (90 days) of combination bicalutamide plus finasteride.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Age ≥ 18 years
3. Eastern cooperative group (ECOG) performance status ≤2
4. Documented histologically confirmed adenocarcinoma of the prostate (minimum 12 core prostate biopsy completed within 90 days of screening)
5. Very low-risk prostate cancer as defined by:

   * Gleason score ≤ 6
   * PSA density ≤ 0.15 ng/mL/mL
   * PSA < 10 ng/mL
   * Clinical tumor stage T1 (cT1) (i.e., no palpable nodule by digital rectal exam)
   * ≤2 prostate cores positive for prostatic adenocarcinoma
   * ≤50% of any given core involved by prostatic adenocarcinoma
6. Willing and qualified for active surveillance at Johns Hopkins
7. Presence of at least one MRI significant visible prostate tumor (i.e., ≥5 mm in at least one dimension) that has been biopsy proven to be prostatic adenocarcinoma Note: MRI may occur pre- or post-prostate biopsy. If done post-biopsy, the MRI must not occur <8 weeks post-prostate biopsy.
8. Serum testosterone ≥150 ng/dL
9. Able to swallow the study drugs whole as a tablet

Exclusion Criteria:

1. Prior local therapy to treat prostate cancer (e.g., radical prostatectomy, radiation therapy, brachytherapy)
2. Prior use of bicalutamide
3. Prior use of finasteride within the past year
4. Prior or ongoing systemic therapy for prostate cancer including, but not limited to:

   * Hormonal therapy (e.g., leuprolide, goserelin, triptorelin)
   * CYP-17 inhibitors (e.g., abiraterone, ketoconazole)
   * Antiandrogens (e.g., bicalutamide, flutamide, nilutamide)
   * Second generation antiandrogens (e.g., enzalutamide, ARN-509)
   * Immunotherapy (e.g., sipuleucel-T, ipilimumab)
   * Chemotherapy (e.g., docetaxel, cabazitaxel)
5. Evidence of serious and/or unstable pre-existing medical, psychiatric or other condition (including laboratory abnormalities) that could interfere with patient safety or provision of informed consent to participate in this study.
6. Any psychological, familial, sociological, or geographical condition that could potentially interfere with compliance with the study protocol and follow-up schedule.
7. Abnormal bone marrow function [absolute neutrophil count (ANC)<1500/mm3, platelet count <100,000/mm3, hemoglobin <9 g/dL]
8. Abnormal liver function (bilirubin, AST, ALT ≥ 3 x upper limit of normal)
9. Abnormal kidney function (serum creatinine ≥ 2 x upper limit of normal)
10. Abnormal cardiac function as manifested by NYHA (New York Heart Association) class III or IV heart failure or history of a prior myocardial infarction (MI) within the last five years prior to enrollment in the study.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Negative re-biopsy rate | three months (90 days)
  To determine the negative re-biopsy rate as determined by MRI/TRUS fusion guided biopsy targeting the dominant nodule site defined by pre-treatment MRI following three months (90 days) of combination bicalutamide plus finasteride.

SECONDARY OUTCOMES:
Rate of exit at 2 years from the active surveillance program at Johns Hopkins due to pathologic upstaging following treatment with bicalutamide plus finasteride. | 2 years
PSA progression rates and PSA progression free survival (PFS), as defined by the Prostate Cancer Working Group 2 (PCWG2) criteria, at 2 years [Scher et al, 2008]. | 2 years
Rate of radiographic disappearance of MRI detectable prostate cancer following treatment with combination bicalutamide plus finasteride (i.e., decrease in size of the target prostate cancer nodule below 5 mm). | 2 years
Adverse events as assessed by the revised National Cancer Institute Common Toxicity Criteria (NCI CTC), version 4.0 published 14 June 2010. | 2 years
Quality of life utilizing the FACT-P and SF36 surveys | 2 years

OTHER OUTCOMES:
Overall rate of exit at 2 years from the active surveillance program at Johns Hopkins following treatment with bicalutamide plus finasteride. | two years
Rate of local treatment (e.g., radical prostatectomy, radiation therapy, brachytherapy) at 2 years and the local treatment free survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Pienta, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States